CLINICAL TRIAL: NCT04663893
Title: Peri-Implant and Peri-Prosthetic Fractures: Epidemiology, Morbility, Mortality, Treatment and Functional Outcome Analysis. A Prospective Multi Center Observational Collaborative Study
Brief Title: Peri-Implant and Peri-Prosthetic Fractures: Epidemiology, Morbidity, Mortality, Treatment and Outcome Analysis
Acronym: PIPPAS
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario 12 de Octubre (Other); Hospital Vall d'Hebron (Other); Hospital de Jove, Gijón, Spain (Unknown); Hospital de Basurto (Other); Hospital Álvaro Cunqueiro (Other); Hospital Galdakao-Usansolo (Other Government); Hospital Universitario de Canarias (Other); Hospital Infanta Elena de Valdemoro, Madrid (Unknown); Hospital Universitario Doctor Peset (Other); Hospital Royo Villanova - Ntra. Sra. de Gracia, Zaragoza (Unknown); Hospital Universitario de Cabueñes, Asturias (Unknown); Hospital Universitario Fundación Alcorcón, Madrid (Unknown); Nuestra Señora de Sonsoles Hospital in Ávila (Other); Hospital Clínico Universitario San Carlos, Madrid (Unknown); Complejo Hospitalario Universitario, A Coruña (Unknown); Hospital Gregorio Marañón, Madrid (Unknown); Hospital Universitario de Álava - Txagorritxu, Alava (Unknown); Hospital Universitario General de Elche, Elche (Unknown); Hospital Gral. Univ. Los Arcos del Mar Menor de Murcia (Unknown); Hospital Vega Baja de Orihuela, Alicante (Unknown); Hospital Gral. Univ. Morales Meseguer, Murcia (Unknown); Hospital Can Misses, Ibiza (Unknown); Hospital Son Llàtzer, Palma de Mallorca (Unknown); Hospital Marqués de Valdecilla, Santander (Unknown); Hospital Virgen de la Salud (Other); Hospital Puerta de Hierro, Madrid (Unknown); Hospital General de Segovia (Other); Hospital Moisés Broggi de Sant Joan Despí, Barcelona (Unknown); Hospital Universitari Sagrat Cor, Barcelona (Unknown); Complejo Hospitalario Llerena-Zafra, Badajoz (Unknown); Hospital Universitario Lucus Augusti (Other); Hospital Universitario La Paz (Other); Hospital Universitario Ramón y Cajal de Madrid (Unknown); Hospital Universitario Pcpe. de Asturias de Alcalá de Henares, Madrid (Unknown); Hospital General Universitario Reina Sofía, Murcia (Unknown); Hospital General Obispo Polanco, Teruel (Unknown); Hospital Universitario de Guadalajara (Unknown); University Hospital of Girona Dr. Josep Trueta (Network); Complejo Hospitalario Universitario de Albacete (Other); Hospital Sierrallana de Torrelavega, Cantabria (Unknown); Complejo Hospitalario de Palencia (Unknown); Hospital Universitario Fundación Jiménez Díaz, Madrid (Unknown); Complexo Hospitalario Universitario de Pontevedra (Unknown); Hospital Parc Taulí de Sabadell, Barcelona (Unknown); Hospital Universitario Miguel Servet, Zaragoza (Unknown); Hospital Universitari Arnau de Vilanova, Lleida (Unknown); Hospital Universitario de León (Unknown); Hospital Universitario de Burgos (Other); Hospital Santa Bárbara, Soria (Unknown); Hospital San Pedro de Logroño (Other); Hospital Costa del Sol de Marbella, Málaga (Unknown); Hospital Parc De Salut Mar, Barcelona (Unknown); Hospital Italiano de Buenos Aires, Argentina (Unknown); Complejo Hospitalario de Navarra (Other); Hospital Santos Reyes de Aranda de Duero, Burgos (Unknown); Hospitales Universitarios Virgen del Rocío (Other); Hospital de la Santa creu i Sant Pau - Barcelona (Other); Hospital Universitario Dr. Negrín, Gran Canaria (Unknown); Hospital Universitario Infanta Leonor, Madrid (Unknown); Hospital Comarcal Alto Guadalquivir de Andújar, Jaén (Unknown); Hospital Universitario de Donostia, Guipúzcoa (Unknown); Hospital Carmen y Severo Ochoa de Cangas de Narcea, Asturias (Unknown); Hospital Reina Sofía de Tudela, Navarra (Unknown); Hospital Universitario San Agustín de Avilés, Asturias (Unknown); Hospital Universitario Virgen de la Macarena, Sevilla (Unknown); Hospital Universitario El Escorial, Madrid (Unknown)
Responsible Party: Principal Investigator, Héctor J Aguado, MD PhD Associate Professor Trauma/Orthogeriatric unit, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 20-2041
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Periprosthetic Fracture of the Upper or Lower Limb; Peri-implant Fracture of the Upper or Lower Limb; Periprosthetic Fractures; Peri-implant Fracture
Keywords: Periprosthetic fracture; peri-implant fracture; mortality; morbidity; loosening; prosthesis revision; fixation; osteosynthesis; complication; ambulate; quality of life
MeSH Terms: conditions — Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study supports Spanish data collection and analysis on Periprosthetic and Peri-implant fractures of the upper and lower limb. Treatment and clinical management of this fractures are complex and goes along with complications. There will be more than 70 hospitals providing information. This study will provide evidence on which is the best treatment for every unique patient. This will help trauma surgeons and geriatricians to provide better treatments, to improve health care in our society, reducing mortality, morbidity, improving functional outcomes, and reducing costs, which in turn will be advances in trauma care.

DETAILED DESCRIPTION:
There is no clinical evidence on which are the best treatment options for Periprosthetic and Peri-implant fractures of the upper and lower limb. This is a multi-center collaborative study seeking to obtain a big number of patients. Data collection includes previous health status and quality of life, which is the clinical management and treatment, as well as the outcome after one month, six months and one year. The investigators will be able to define risk factors and clinical attitudes, which influence on the patient outcome. And therefore, be able to establish treatment protocols and give management recommendations based on the observed clinical evidence to improve healing indexes, morbidity and mortality, function, grade of autonomy and quality of live.

Main questions to be answered are: 1. which is the epidemiology of Periprosthetic and Peri-implant fractures and how are they treated in Spain, 2. Identify risk factors for complications and worse outcomes, 3. which is the morbidity and mortality, 4. influence of the fracture type and implants already placed on management and outcome, 5. influence of the treatment on patients' grade of independency, and 6. identified which are the risk factors for treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the diagnose of Periprosthetic fracture of the shoulder, elbow, hip or knee. Or patients with the diagnose of Peri-implant fracture of the scapula, humerus, forearm, pelvis, femur, patella, tibia or fibula. Or patient presenting cut-out or cut-in after DHS or nail after a proximal humeral fracture.
* 18 years or older

Exclusion Criteria:

* Spine PP or PI fracture
* PP or PI secondary to metastasis or tumoral fracture
* PP or PI intraoperative fracture
* PP or PI pathologic fracture
* PP ankle fracture
* PP or PI wrist or hand fracture
* Fixation failure without any new fracture line: except cut-out or cut-in after DHS or nail of a proximal humeral fracture.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for a Periprosthetic or a Peri-implant fracture of the upper or lower limb by any participant hospital in Spain.
  Hospital participation is voluntary and upon request or invitation. 80 hospitals participating all over Spain
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 12 months
  Rate of mortality at anytime from fracture diagnose up to 12 months
Fracture classification | Pre-operatively (Day -1)
  Fracture classification using the UCS for periprosthetic fractures, and the adapted H. Broggi classification for peri-implant fractures. Number of patients in each classification group
Treatment | Post-operatively (Day +1)
  Number of patients treated with fixation or revision and fixation or implant removal

SECONDARY OUTCOMES:
Fracture healing | Up to 12 months
  Rate of bone union on X-rays
Health related quality of life | Up to 12 months
  EuroQuality of Life 5Dimensions 5Leves (EQ5D5L)
Dependency | Up to 12 months
  Clinical frailty scale (1-9) 1=very fit, 9=terminally ill
Mental situation | Up to 12 months
  Pfeiffer test
Gait | Up to 12 months
  FFN-MCD mobility scale (Fragility Fracture Network-Minimum Common Dataset). 1-5: 1=independent mobility, 5=No functional mobility
Bone protector treatment | Up to 12 months
  Is the patient under treatment with vitamine D, calcium, bone formation, bone modeling?
Life style change | Up to 12 months
  Need to change place of living because of the fracture or its sequels.
Medical or Surgical complications | Up to 12 months
  in need of at least one in-hospital night.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor J Aguado, MD PhD, Study Director — Hospital Clínico Universitario Valladolid; Pablo Castillón, MD PhD, Study Director — Mútua Universitaria de Terrassa; Josep M Muñoz Vives, MD PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa; Cristina Ojeda-Thies, MD PhD, Principal Investigator — Hospital 12 de Octubre, Madrid; Pilar Camacho, MD PhD, Principal Investigator — Hospital Clinic of Barcelona; Jordi Teixidor, MD, Principal Investigator — Hospital Universitario Vall d´Hebrón; Pablo García-Portablella, MD, Principal Investigator — Hospital de Jove, Gijón
Locations (7):
- Spain (7):
  - Mutua Universitaria de Tarrasa, Barcelona
  - Althaia, Xarxa Assistencial Universitària de Manresa, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - Hospital de Jove, Gijón
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 1st of January 2022
Access Criteria: Application form to the PIPPAS study office. The applicant must be a study participant and should describe which is the substudy to be held, providing a detailed description and variables need for that reason.

REFERENCES:
- [Derived] Moreta J, Aguado HJ, Castillon-Bernal P, Munoz-Vives JM, Camacho P, Jornet-Gibert M, Teixidor J, Pereda-Manso A, Garcia-Sanchez Y, Ojeda-Thies C, Garcia-Portabella P, Alvarez EM, Noriega-Gonzalez D, Munoz-Moreno MF, Arroyo-Hernantes I, Alvarez-Ramos BA, Garcia-Medrano B, Martinez-Selles C, Marin-Jimenez S, Garcia-Virto V, Pais-Ortega S, Acha A, Tomas-Hernandez J, Selga-Marsa J, Andres-Peiro JV, Piedra-Calle C, Blasco-Casado F, Guerra-Farfan E, Querolt-Coll J, de Santamaria GT, Hernandez JM, Renau-Cerrillo M, Gil-Aliberas C, Carreras-Castaner A, Vives-Barquiel M, Fernandez EA, Manzano EF, De Cortazar UG, Arrieta M, Escobar D, Castrillo E, Balvis Balvis P, Denisiuk M, Menendez MC, Pastor S, Larrazabal A, Olias-Lopez B, Amaya-Espinosa P, Boluda-Mengod J, Gonzalez-Martin D, Lopez-Dorado D, Borras-Cebrian JC, Martinez-Perez C, Pazmino PAF, Calavia-Cale P, Suarez-Suarez MA, Lanuza-Lagunilla L, Arias AG, Cabria-Fernandez J, Garcia-Coiradas J, Valle-Cruz J, Del Saz JS, Mora-Fernandez J, Lalueza-Andreu P, Bonome-Roel C, Cano-Leira MA, Carrasco AB, Pariza AL, Fernandez-Juan A, la Puente CS, Juldain-Mondragon M, Arsuaga JG, Saura-Sanchez E, Gimenez-Ibanez S, Sanchez-Gomez P, Ricon-Recarey FJ, Garcia Garcia EM, Cuadrado-Abajo F, Perez-Nunez MI, Del Pozo-Manrique P, Navas-Garcia FMG, Garcia-Paredero E, Guijarro-Valtuena A, Robles TB, Navas-Pernia I, De Villasante-Jiron I, Porta TS, Becerra CC, Otero-Naveiro V, Paz SP, Castrillo IF, Fernandez-Dorado F, Martinez-Menduina A, Vaquerizo-Garcia V, Murcia-Asensio A, Galian-Munoz E, Marin-Martinez C, Munoz-Vicente A, Plaza-Salazar N, Gamez-Asuncion C, Benito-Santamaria J, Salgado-Tarrida P, Prats-Puente O, Cuenca-Copete A, Gonzalez-Montero B, Giraldo-Vegas LA, Mingo-Robinet J, Briso-Montiano R, Barberia-Biurrun A, Escudero-Martinez E, Chouza-Montero L, Naharro-Tobio M, Gasset-Teixidor A, Dominguez-Ibarrola A, Penalver JM, Serrano-Sanz J, Roche-Albero A, Martin-Hernandez C, Macho-Mier M, Salo-Cuenca JC, Rosello JE, Criado-Albillos G, Cabello-Benavides HG, Nestar DA, Gonzalez-Bernal J, Gonzalez-Santos J, Cunchillos-Pascual J, Blasco JM, Bogallo-Dorado JM, Ramirez-Roldan A, Cano-Porras JR, Marques-Lopez F, Martinez-Diaz S, Slullitel PI, Carabelli GS, Astore I, Boietti BR, Cordova-Peralta JC, Hernandez-Pascual C, Rodriguez-Gangoso A, Dot-Pascuet I, Pineiro-Borrero A, Perez-Sanchez JM, Mandia-Martinez A, De Caso-Rodriguez J, Martin-Marcuello J, Benito-Mateo M, Alda-Gastiain O, Corcuera-Elosegui I, Gonzalez-Panisello MR, Perez-Salazar NE, De Sande-Diaz M. Internal fixation versus revision arthroplasty for Vancouver B2-B3 fractures: mortality and functional outcomes in frail patients. Insights from the PIPPAS study of 485 patients. J Orthop Traumatol. 2025 Dec 22;26(1):78. doi: 10.1186/s10195-025-00886-3. PMID 41428314
- [Derived] PIPPAS Study Group. Optimizing periprosthetic fracture management and in-hospital outcome: insights from the PIPPAS multicentric study of 1387 cases in Spain. J Orthop Traumatol. 2024 Mar 7;25(1):13. doi: 10.1186/s10195-024-00746-6. PMID 38451303